CLINICAL TRIAL: NCT06084416
Title: A Phase 1b Dose Optimization Study of Sovilnesib (an Oral KIF18A Inhibitor) in Subjects With Advanced High Grade Serous Ovarian Cancer
Brief Title: A Study of Sovilnesib in Subjects With Ovarian Cancer
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Volastra Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SOVI-2302
Record Dates: First submitted 2023-10-10; First posted 2023-10-16 (Actual); Last update posted 2025-10-20 (Actual); Status verified 2025-10

CONDITIONS: High Grade Serous Adenocarcinoma of Ovary; Fallopian Tube Cancer; Primary Peritoneal Carcinoma; Chromosomal Instability
Keywords: KIF18A Inhibitor
MeSH Terms: conditions — Fallopian Tube Neoplasms; Chromosomal Instability

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (4):
- Dose Level 1 (Experimental): Subjects will receive sovilnesib once daily at Dose Level 1 in 28-day cycles.
  Interventions: Drug: Sovilnesib
- Dose Level 2 (Experimental): Subjects will receive sovilnesib once daily at Dose Level 2 in 28-day cycles.
  Interventions: Drug: Sovilnesib
- Dose Level 3 (Experimental): Subjects will receive sovilnesib once daily at Dose Level 3 in 28-day cycles.
  Interventions: Drug: Sovilnesib
- Dose Level 4 (Experimental): Subjects will receive sovilnesib once daily at Dose Level 4 in 28-day cycles.
  Interventions: Drug: Sovilnesib

INTERVENTIONS:
Drug: Sovilnesib — Sovilnesib tablets will be given orally.

SUMMARY:
This is a randomized, phase 1b study to assess the safety, tolerability, pharmacokinetics (PK), and efficacy of sovilnesib at different dose levels to establish the Recommended Phase 2 Dose (RP2D) of sovilnesib in subjects with high grade serous ovarian cancer (HGSOC).

DETAILED DESCRIPTION:
This is a randomized, phase 1b dose optimization study of sovilnesib in subjects with platinum-resistant HGSOC. The focus of the proposed clinical study is to establish the RP2D of sovilnesib in HGSOC.

An adaptive multi-cohort design will be used to assess the safety, tolerability, PK, and efficacy of multiple dose levels in parallel to establish the RP2D of sovilnesib. The study will be conducted in 2 parts.

Part 1: 10 subjects will be randomized to each of the open dose levels to generate preliminary PK, pharmacodynamic (PD), safety, tolerability and efficacy data. Early stopping rules for safety based on a Bayesian Toxicity Monitoring Design will be applied.

Part 2: Based on review of the data from Part 1, 20-30 additional subjects will be randomized to 2 or more dose levels examined in Part 1. At the end of Part 2, PK, PD, safety, tolerability and efficacy data will be used to determine the RP2D. Early stopping rules for safety based on a Bayesian Toxicity Monitoring Design and for futility based on a Bayesian Efficacy Monitoring via Predictive Probability Design will be applied.

Sovilnesib will be given orally in 28-day cycles at selected dose levels of interest. Dosing will continue until disease progression, unacceptable toxicity, withdrawal of consent, or other stopping criteria are met.

ELIGIBILITY:
Key Inclusion Criteria:

* All Parts: Age ≥ 18 years, ECOG Performance Status ≤ 1, at least 1 site of measurable disease evaluable by CT scan or MRI per RECIST 1.1, able to take oral medication without alteration
* High Grade Serous Ovarian Cancer, Fallopian Tube or Primary Peritoneal Cancer - histologically or cytologically confirmed; metastatic or unresectable; platinum resistant (defined as recurrence within 6 months of platinum containing therapy) or platinum refractory; prior bevacizumab treatment, or ineligible or intolerant to bevacizumab, or did not receive bevacizumab based on Investigator judgement; if germline and/or somatic BRCA1/2 mutation, previously treated with PARP-inhibitor or ineligible or intolerant.

Key Exclusion Criteria:

* MSI-H, dMMR, POLE gene hotspot mutated, or known hypermutator phenotype
* Endometrioid, clear cell, mucinous, sarcomatoid, low-grade/borderline ovarian tumor or mixed tumors containing any of the above histologies
* Previously received KIF18A inhibitor
* Current CNS metastases or leptomeningeal disease
* Cardiac parameters: MI or stroke ≤ 6 months, unstable angina/PE/DVT/CABG ≤ 6 months, NYHA Class ≥ II, LVEF < 50%
* Any gastrointestinal condition (e.g. malabsorption syndrome, surgical anastomosis, short bowel syndrome) that might affect the absorption of oral medications including the study drug

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 120 (Estimated)
Dates: Start 2024-04-04 (Actual); Primary Completion 2026-03 (Estimated); Study Completion 2026-04 (Estimated)

PRIMARY OUTCOMES:
Determination of the Recommended Phase 2 Dose (RP2D) of Sovilnesib | Up to 24 months
Frequency and duration of Serious Adverse Events (SAEs) graded according to the National Cancer Institute Common Terminology Criteria for Adverse Events (NCI-CTCAE) version 5.0 | Up to 24 months
Frequency and duration of Treatment-related Adverse Events (AEs) graded per NCI-CTCAE version 5.0 | Up to 24 months
Frequency and duration of Treatment-Emergent AEs (TEAEs) graded per NCI-CTCAE version 5.0 | Up to 24 months
Frequency of Dose Interruptions and Permanent Treatment Discontinuations | Up to 24 months
Objective Response Rate (ORR) as assessed by Response Evaluation Criteria in Solid Tumors (RECIST) version 1.1 | Up to 24 months

SECONDARY OUTCOMES:
Duration of Response (DOR) as assessed by RECIST version 1.1 | Up to 24 months
Disease Control Rate (DCR) as assessed by RECIST version 1.1 | Up to 24 months
Progression Free Survival (PFS) as assessed by RECIST version 1.1 | Up to 24 months
Evaluation of CA-125 response by Gynecologic Cancer InterGroup (GCIG) criteria | Up to 24 months
Plasma level of Sovilnesib | Up to 24 months

CONTACTS AND LOCATIONS:
Locations (13):
- United States (13):
  - The University of Alabama at Birmingham, Birmingham, Alabama
  - University of Arkansas for Medical Sciences, Little Rock, Arkansas
  - UCLA, Los Angeles, California
  - Hoag Memorial Hospital, Newport Beach, California
  - Georgia Cancer Center Augusta University, Atlanta, Georgia
  - Johns Hopkins Hospital, Baltimore, Maryland
  - Dana Farber Cancer Institute, Boston, Massachusetts
  - Corewell Health, Grand Rapids, Michigan
  - Roswell Park Comprehensive Cancer Center, Buffalo, New York
  - Icahn School of Medicine at Mount Sinai, New York, New York
  - OU Health Stephenson Cancer Center, Oklahoma City, Oklahoma
  - MUSC Hollings Cancer Center, Charleston, South Carolina
  - Fred Hutchinson Cancer Center, Seattle, Washington

IPD SHARING:
Plan to Share IPD: Undecided